CLINICAL TRIAL: NCT00267501
Title: Eosinophils and Inflammation, an Expanded Study
Brief Title: Data and Sample Collection Study to Elucidate the Mechanisms of Eosinophilic Disorders
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 04-12-8 : 2008-0090; R01 DK075401
Record Dates: First submitted 2005-12-15; First posted 2005-12-21 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Eosinophilic Gastrointestinal Disease Eosinophilic Inflammatory Disease; Food Allergy
Keywords: Eosinophilic Disorders
MeSH Terms: conditions — Food Hypersensitivity; Eosinophilia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The purpose of this study is to elucidate the mechanisms underlying eosinophil growth, survival, migration, and function and to investigate and further characterize the pathophysiology of, clinical manifestations of, and spectrum of disease severity of eosinophilic inflammation in humans.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from the patient or parent/guardian. Assent will be obtained from all minors 11 years of age and older.
* Carrying a diagnosis of eosinophilic gastrointestinal disease, eosinophilic inflammatory disease, or food allergy OR family member, or normal control

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with eosinophilic disorders and patients without eosinophilic disorders to serve as normal controls
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-05; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, M.D., Ph.D., Principal Investigator — Cincinnati Children's Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States